CLINICAL TRIAL: NCT03289767
Title: Simple Preparation of Endotracheal Tube for Optimal Angulation During Intubation: A Randomized Controlled Trial
Brief Title: Simple Preparation of Endotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: JHSeo_angulation
Record Dates: First submitted 2017-09-12; First posted 2017-09-21 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Endotracheal Tube

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curved-tube (Experimental): Giving additional curve to the endotracheal tube by simple preparation.
  Interventions: Other: Curved-tube
- Control (No Intervention): No other manipulation of the endotracheal tube is done.

INTERVENTIONS:
Other: Curved-tube — Connecting both ends of the endotracheal tube ("O" shape) for 5-min and releasing it provides additional anterior angle temporarily.
  Arms: Curved-tube

SUMMARY:
To observe the effect of additional E-tube angulation on intubation time and success rate.

DETAILED DESCRIPTION:
The hypothesis of this study is that shaping endotracheal tube by end-to-end connection before induction will provide more optimal angulation for endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective surgery requiring general anesthesia and tracheal intubation

Exclusion Criteria:

* Patients with congenital or acquired upper airway lesions
* Patients with high risk of aspiration

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Successful intubation on first attempt | On endotracheal intubation up to 1 min
  Whether successful intubation is done on first attempt or on additional attempt

SECONDARY OUTCOMES:
Time to intubate (TIT) | On endotracheal intubation up to 1 min
  The TIT started when the blade first passed the lips, and ended when the the detection of end-tidal CO2 trace

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwa Seo, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea